CLINICAL TRIAL: NCT05809674
Title: Polarization Sensitive Optical Coherence Tomography - Phase II: A Pilot Study
Brief Title: Polarization Sensitive Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: R1819/61/2021
Record Dates: First submitted 2023-02-12; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult Cohort: * Aged 21 and above
  * Ability to provide informed consent
  * 42 normal controls: No diabetes and free from clinically relevant eye disease that interferes with the aim of the study i.e. glaucoma, diabetic retinopathy, age-related macular degeneration, uveitis, or vascular occlusive diseases
  * 76 subjects with pathological myopia (up to -12 dioptres) or staphyloma
  Interventions: Device: Polarization sensitive optical coherence tomography (PS-OCT)
- Children Cohort: * Aged 10 to 18
  * 23 subjects with low to moderate myopia (-0.75 to -6 dioptres)
  * 23 subjects with high myopia (more than -6 dioptres)
  * Ability of legal representative and subject to provide informed consent
  Interventions: Device: Polarization sensitive optical coherence tomography (PS-OCT)

INTERVENTIONS:
Device: Polarization sensitive optical coherence tomography (PS-OCT) — The PS-OCT is a prototype, also known as an early version of a medical device, specially developed by the Ocular Imaging Research Group, Singapore Eye Research Institute, for prediction of myopia progression. It has not been approved for use in any other country. There is currently no method to identify who is at risk of myopia progression. The PS-OCT device will provide the capabilities of OCT scleral biomarkers, which may have the potential to identify individuals at high risk for myopia.

SUMMARY:
The purpose of the study is to use the polarization sensitive optical coherence tomography (PS-OCT) developed by Singapore Eye Research Institute, to evaluate the potential OCT scleral biomarkers capable of predicting risk of myopia progression.

ELIGIBILITY:
Inclusion Criteria:

(Adult Cohort)

* Aged 21 and above
* Ability to provide informed consent
* 42 normal controls: No diabetes and free from clinically relevant eye disease that interferes with the aim of the study i.e. glaucoma, diabetic retinopathy, age-related macular degeneration, uveitis, or vascular occlusive diseases
* 76 subjects with pathological myopia (up to -12 dioptres) or staphyloma

(Children Cohort)

* Aged 10 to 18
* 23 subjects with low to moderate myopia (-0.75 to -6 dioptres)
* 23 subjects with high myopia (more than -6 dioptres)
* Ability of legal representative and subject to provide informed consent

Exclusion Criteria:

(Adult Cohort)

* Unable to give consent
* Subjects with visual acuity worse than 6/12
* Diagnosis of clinically relevant eye disease that interferes with the aim of the study (e.g. diabetic retinopathy, hereditary macular disease, glaucoma, uveitis, or vascular occlusive diseases) or conditions that may potentially result in poor quality imaging scans (severe cataract, corneal haze/opacity)

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and children cohorts
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Primary Aim | 1.5 years
  High reproducibility in myopia cases as shown in PS-OCT derived sclera anisotropy patterns

SECONDARY OUTCOMES:
Secondary Aim | 1.5 years
  Changes in scleral anisotropy in adults with different degrees of myopia (up to -12 dioptres), as associated with the presence of staphyloma

OTHER OUTCOMES:
Tertiary Aim | 1.5 years
  Anisotropy correlation with refraction and axial length in children with low (-0.75 to -6 dioptres) and high (more than -6 dioptres) myopia, as measured by PS-OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore